CLINICAL TRIAL: NCT05884437
Title: The Effects of Chiropractic Care on the Brain, Autonomic Nervous System, Gait, and Patient Reported Outcomes in Adults With Diagnosed or Suspected Metabolic Syndrome: a Proof-of-concept Trial
Brief Title: The Effects of Chiropractic in Adults With Metabolic Syndrome
Acronym: MET
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Prioritizing other studies
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: I-0023
Record Dates: First submitted 2023-02-16; First posted 2023-06-01 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Syndrome
Keywords: Chiropractic; Metabolic syndrome; Spinal manipulation; autonomic nervous system; EEG; patient reported outcomes
MeSH Terms: conditions — Metabolic Syndrome | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: Single-arm pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chiropractic (Experimental): Chiropractic adjustment
  Interventions: Procedure: Chiropractic adjustment

INTERVENTIONS:
Procedure: Chiropractic adjustment — Participants will receive 6 weeks of chiropractic care. The frequency of care will be determined by the field clinician. Participants will have their spine assessed for the presence of vertebral subluxations per their clinician's normal and customary procedures. The adjustment technique(s) utilized by the field clinician will be at their discretion.

SUMMARY:
The purpose of this study is to assess the feasibility of our study procedures/protocols and to look at the potential effects of chiropractic care on people with metabolic syndrome.

DETAILED DESCRIPTION:
After providing informed consent, individuals will undergo 6 weeks of chiropractic care. Throughout these 6 weeks there will be three assessments (Day 0, Week 2, and Week 6) that each include the following:

1. Seated resting recording
2. Auditory oddball task
3. Isometric hand grip
4. Postural challenge
5. Treadmill walking
6. Patient-reported outcome surveys

Each assessment will consist of the following recordings:

1. Electroencephalography [EEG]
2. Electrodermal activity [EDA]
3. Impedance cardiography [ICG]
4. Electrocardiogram [ECG]

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 18
* Individuals who can wear an EEG net for 30 minutes
* Individuals who can sit quietly for at least 15 minutes
* Individuals who can walk unassisted for up to 10 minutes
* Individuals who can provide informed consent
* Individuals who meet 3 of the 5 following criteria:

  * Elevated waist circumference (>40 in/102 cm if male and >35 in/88cm if female)
  * Elevated triglycerides (>150 mg/dL) or drug treatment for elevated triglycerides
  * Reduced HDL-cholesterol (<40mg/dL if male and <50 mg/dL if female) or drug treatment to increase HDL-C
  * Elevated blood pressure (>130 mm Hg systolic BP or >85 mm Hg diastolic BP) or drug treatment to reduce blood pressure
  * Elevated fasting glucose (>100 mg/dL) or drug treatment to reduce blood glucose

Exclusion Criteria:

* Individuals with a known disorder resulting in syncope/fainting during postural changes (e.g., POTS, orthostatic hypotension)
* Individuals with impaired function of the dominant hand
* Individuals with malignant hypertension
* Individuals with a known heart condition such as arrhythmia that results in an aberrant ECG recording
* Individuals with any implanted devices (i.e., pacemakers)
* Individuals with brain aneurysms
* Individuals with a history of epilepsy or stroke that would influence EEG readings
* Individuals with a diagnosed externalizing or thought disorder (i.e., anti-social disorder, any major personality disorder such as borderline personality disorder, or schizophrenia)
* Individuals who are on short-acting benzodiazepines which include midazolam & triazolam
* Individuals with any serious injury or surgery to the head or torso, or lower body in the last 6 months
* Individuals with a hearing impairment or hearing aids (due to the auditory stimulus recording being performed)
* Individuals who are currently pregnant
* Individuals with current litigation related to a physical, health-related injury
* Individuals who have been diagnosed with rheumatoid arthritis, osteoporosis or instability of the neck.
* Individuals with moderate to severe pain on a daily basis
* Pain on the day of testing rated greater than 3/10 on a visual analog scale (VAS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | through study completion, an average of 1 year
  Length of time needed to recruit target number of participants
Participant adherence rate | through study completion, an average of 1 year
  Proportion of participants able to adhere to the testing & treatment schedule
Participant tolerability rate | through study completion, an average of 1 year
  Proportion of participants able to perform all aspects of the testing regimen
Participant retention rate | through study completion, an average of 1 year
  Proportion of enrolled participants who complete the full testing regimen
Acceptability of treatment regimen for participants | Week 6
  9-item acceptability questionnaire

SECONDARY OUTCOMES:
EEG resting state broadband power | Day 1
  64-channel hydronet cap
EEG resting state broadband power | Week 2
  64-channel hydronet cap
EEG resting state broadband power | Week 6
  64-channel hydronet cap
EEG resting state functional connectivity | Day 1
  64-channel hydronet cap
EEG resting state functional connectivity | Week 2
  64-channel hydronet cap
EEG resting state functional connectivity | Week 6
  64-channel hydronet cap
EEG evoked latency | Day 1
  64-channel hydronet cap during auditory oddball task
EEG evoked latency | Week 2
  64-channel hydronet cap during auditory oddball task
EEG evoked latency | Week 6
  64-channel hydronet cap during auditory oddball task
EEG evoked amplitude | Day 1
  64-channel hydronet cap during auditory oddball task
EEG evoked amplitude | Week 2
  64-channel hydronet cap during auditory oddball task
EEG evoked amplitude | Week 6
  64-channel hydronet cap during auditory oddball task
skin conductance level (SCL) | Day 1
  2 electrodermal activity (EDA) sensors on first and second digits of non-dominant hand
skin conductance level (SCL) | Week 2
  2 electrodermal activity (EDA) sensors on first and second digits of non-dominant hand
skin conductance level (SCL) | Week 6
  2 electrodermal activity (EDA) sensors on first and second digits of non-dominant hand
Impedance cardiogram (ICG) pre-ejection period (PEP) | Day 1
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) pre-ejection period (PEP) | Week 2
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) pre-ejection period (PEP) | Week 6
  2 sensors on chest and 2 sensors on back
ECG mean interbeat interval | Day 1
  3 sensors on torso
ECG mean interbeat interval | Week 2
  3 sensors on torso
ECG mean interbeat interval | Week 6
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | Day 1
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | Week 2
  3 sensors on torso
ECG respiratory sinus arrhythmia (RSA) | Week 6
  3 sensors on torso
ECG de-trended fluctuation analysis | Day 1
  3 sensors on torso
ECG de-trended fluctuation analysis | Week 2
  3 sensors on torso
ECG de-trended fluctuation analysis | Week 6
  3 sensors on torso
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | Day 1
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | Week 2
  2 sensors on chest and 2 sensors on back
Impedance cardiogram (ICG) initial systolic time interval (ISTI) | Week 6
  2 sensors on chest and 2 sensors on back
Electrodermal activity (EDA) non-specific skin conductance responses (SCR) | Day 1
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) non-specific skin conductance responses (SCR) | Week 2
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) non-specific skin conductance responses (SCR) | Week 6
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) power spectral density (PSD) | Day 1
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) power spectral density (PSD) | Week 2
  2 sensors on first and second digits of non-dominant hand
Electrodermal activity (EDA) power spectral density (PSD) | Week 6
  2 sensors on first and second digits of non-dominant hand
Composite Autonomic Symptom Score (COMPASS-31) | Day 0
  31-item questionnaire
Composite Autonomic Symptom Score COMPASS-31) | Day 1
  31-item questionnaire
Composite Autonomic Symptom Score (COMPASS-31) | Week 2
  31-item questionnaire
Composite Autonomic Symptom Score (COMPASS-31) | Week 6
  31-item questionnaire
Patient-Reported Outcomes Measurement Information System Cognitive Abilities and Cognitive Concerns Scale (PROMIS-Cog) | Day 0
  8-item questionnaire
Patient-Reported Outcomes Measurement Information System Cognitive Abilities and Cognitive Concerns Scale (PROMIS-Cog) | Day 1
  8-item questionnaire
Patient-Reported Outcomes Measurement Information System Cognitive Abilities and Cognitive Concerns Scale (PROMIS-Cog) | Week 2
  8-item questionnaire
Patient-Reported Outcomes Measurement Information System Cognitive Abilities and Cognitive Concerns Scale (PROMIS-Cog) | Week 6
  8-item questionnaire
Perceived Stress Scale (PSS) | Day 0
  10-item questionnaire
Perceived Stress Scale (PSS) | Day 1
  10-item questionnaire
Perceived Stress Scale (PSS) | Week 2
  10-item questionnaire
Perceived Stress Scale (PSS) | Week 6
  10-item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tyson Perez, DC, PhD, Principal Investigator — Life University
Locations (1):
- Dr. Sid E. Williams Center for Chiropractic Research, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No